CLINICAL TRIAL: NCT04244448
Title: A Study of Bioequivalence When Administering Biktarvy® (TAF/FTC/BIC) in the Form of a Solid/Crushed/Dissolved Tablet to Healthy Volunteers - SOLUBIC Study
Brief Title: Bioequivalence of Solid/Crushed/Dissolved Forms of Biktarvy®
Acronym: SOLUBIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-211
Record Dates: First submitted 2019-12-12; First posted 2020-01-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BIKTARVY® ADMINISTRATION DISSOLVED IN WATER (Other): BIKTARVY® route in healthy volunteers: dissolved in water in Pharmacokinetics study protocol Compare the pharmacokinetic (PK) of dissolved in water versus crushed and solid form of BIKTARVY® in the same healthy volunteer, to determine if there is a PK equivalence between these three modes of administration of BIKTARVY®.
  Interventions: Drug: receive dissolved form of BIKTARVY®
- BIKTARVY® ADMINISTRATION CRUSHED (Other): BIKTARVY® route in healthy volunteers: crushed in Pharmacokinetics study protocol Compare the pharmacokinetic (PK) of crushed versus dissolved in water and solid form of BIKTARVY® in the same healthy volunteer, to determine if there is a PK equivalence between these three modes of administration of BIKTARVY®.
  Interventions: Drug: receive crushed form of BIKTARVY®
- BIKTARVY® ADMINISTRATION SOLID (Other): BIKTARVY® route in healthy volunteers: solid tablet in Pharmacokinetics study protocol Compare the pharmacokinetic (PK) of solid form of BIKTARVY® versus dissolved in water and crushed in the same healthy volunteer, to determine if there is a PK equivalence between these three modes of administration of BIKTARVY®.
  Interventions: Drug: receive solid form of BIKTARVY®

INTERVENTIONS:
Drug: receive dissolved form of BIKTARVY® — The healthy volunteers will receive dissolved form of BIKTARVY® Pharmacokinetic samples will be taken at the following times: 0 hour (right before taking Biktarvy®); 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 8 hours; 12 hours; 24 hours; 36 hours; 48 hours and 72 hours (after Biktarvy®).
  Other Names: no other intervention name
  Arms: BIKTARVY® ADMINISTRATION DISSOLVED IN WATER
Drug: receive crushed form of BIKTARVY® — The healthy volunteers will receive crushed form of BIKTARVY® Pharmacokinetic samples will be taken at the following times: 0 hour (right before taking Biktarvy®); 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 8 hours; 12 hours; 24 hours; 36 hours; 48 hours and 72 hours (after Biktarvy®).
  Other Names: no other intervention name
  Arms: BIKTARVY® ADMINISTRATION CRUSHED
Drug: receive solid form of BIKTARVY® — The healthy volunteers will receive solid form of BIKTARVY® Pharmacokinetic samples will be taken at the following times: 0 hour (right before taking Biktarvy®); 0.5 hour; 1 hour; 1.5 hours; 2 hours; 2.5 hours; 3 hours; 4 hours; 8 hours; 12 hours; 24 hours; 36 hours; 48 hours and 72 hours (after Biktarvy®).
  Other Names: no other intervention name
  Arms: BIKTARVY® ADMINISTRATION SOLID

SUMMARY:
Study context:

Some HIV-positive patients have difficulties with oral administration of antiretroviral drugs, such as children and adults suffering from ENT cancer. It is therefore necessary to offer these patients an alternative: administering the triple therapy in a liquid or well crushed form would be alternatives to a solid tablet, conditional on demonstrating their bioequivalence and that they are well tolerated (taste in particular).

Objectives:

The investigator's primary intention is to demonstrate the bioequivalence of each of the three active ingredients in Biktarvy® (single daily tablet made up of a set combination of tenofovir alafenamide/emtricitabine/bictegravir: TAF/FTC/BIC) by administering the drug in the forms of a complete and solid tablet (phase S), a tablet dissolved in water (phase D) or a tablet crushed and suspended in apple compote (phase C). The secondary objectives are to compare the safety, tolerance (taste in particular) and preference of healthy volunteers after administration of Biktarvy®, depending on the three methods of oral administration.

Equipment and methods:

This is a phase I, monocentric, open, three-period, randomised, cross-over trial that will be conducted with 18 healthy volunteers (9 men, 9 women) above the age of 18 in a French university hospital (Caen University Hospital - CHU de Caen). The healthy volunteers will be randomised to receive three different forms (solid, dissolved or crushed) in a varying order, according to the randomisation, at an interval of 14 to 28 days. After each of the three doses, the volunteers will be hospitalised for 24 hours and will then return three times to carry out the pharmacokinetic study with samples taken at the following times: 0 h (right before taking Biktarvy®); 0.5 h; 1 h; 1.5 h; 2 h; 2.5 h; 3 h; 4 h; 8 h; 12 h; 24 h; 36 h; 48 h and 72 h (after Biktarvy®).

The plasma concentration in antiretroviral drugs will be analysed by liquid chromatography-mass spectrometry (QTRAP 5500, Sciex, Les Ulis, France) at Orléans Regional Hospital (CHR d'Orléans). The bioequivalence between administration methods D or C will be demonstrated if the confidence interval at 90% (CI 90%) of the ratio parameters Cmax, AUC0-72h and AUC0-∞ is included in the 80%-125% range of those obtained for administration method S and for the three active ingredients.

Hypothesis tested:

Oral administration of Biktarvy® tablets dissolved in water (as a liquid solution) or crushed and administered in an apple compote is bioequivalent to the solid form (entire tablet swallowed with water) with regard to the three active ingredients that make up Biktarvy®. This means that these methods could be offered to patients who have difficulties with swallowing tablets. Preliminary data must be obtained using healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 18 and 55 years old, confirmed as being in good health by an attending physician based on a medical evaluation that includes medical history, taking vital signs, a physical examination, clinical laboratory tests and an ECG.
* Subject does not present any intolerance or anterior skin rashes under the study drugs (TAF, FTC, BIC).
* Subject has a body mass index of between 18 and 30 kg/m2, inclusive.
* Subject's test results are negative for HIV and Hepatitis B and C.
* Subject's veins are in good condition.
* Non-smoking subject who has not consumed nicotine or products containing nicotine for 90 days before taking the first treatment in the study.
* Participant is part of a social security scheme.
* Subject is able and willing to sign the informed consent form before the preliminary evaluations.

Exclusion Criteria:

* Subject's creatinine clearance is below 50 mL/min.
* Pregnant or breastfeeding women.
* Women of reproductive age without adequate contraception, such as: contraceptive pill, hysterectomy, sterilisation, intra-uterine device (coil), total abstinence, dual methods of contraception or two years after menopause. Women must agree to take precautions to avoid becoming pregnant for the duration of the study.
* Men in a relationship without adequate contraception.
* Subject taking any treatment (during the two weeks before Day 1) that could interfere with the study medications (TAF, FTC, BIC): rifampicin, St. John's wort, antacids containing magnesium and/or aluminium, iron-based drugs, carbamazepine, ciclosporin, oxcarbazepine, phenobarbital, phenytoin, rifabutin, rifapentine, sucralfate, macrolides, verapamil, dronedarone, metformin, antimycobacterial medications, antifungal medications, supplements containing calcium, sertraline or methadone.
* Subject with a relevant medical history or current illnesses that are likely to interfere with the absorption, distribution, metabolism or excretion of the medication.
* Subjects with liver enzyme rates (ALAT, ASAT) of alkaline phosphatase and bilirubin higher than or equal to 1.5 times the upper normal value.
* Albumin <35 g/L, serum total protein <65 g/L
* Subject has a QTc <450 ms
* Subject with a pre-existing condition, a surgical sequela or a medical device that disrupts normal gastro-intestinal anatomy or motility or liver and/or kidney function, damaging the absorption, metabolism and/or excretion of the study drugs. A subject who has a medical history of a cholecystectomy, peptic ulcers, inflammatory intestinal diseases or pancreatitis must be excluded.
* Subject has a history of drug, alcohol or solvent abuse or currently abuses such substances.
* Subject is under guardianship or trusteeship.
* Subject is unable to understand the nature and scope of the study and the required procedures.
* Subject who participated in a study with the medication in the 60 days before the first day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of each of the three active ingredients in Biktarvy® | 0 - 72 hours
  Measurement of plasma concentration of each of the three active ingredients in Biktarvy® (TAF/FTC/BIC), administered in the forms of a complete and solid tablet (phase S), a tablet dissolved in water (phase D) or a tablet crushed and suspended in apple compote (phase C)
  Samples taken at the following times:
  0 hour (right before taking Biktarvy®); 0.5 hour; 1 hours; 1.5 hour; 2 hours; 2.5 hours; 3 hours; 4 hours; 8 hours; 12 hours; 24 hours; 36 hours; 48 hours and 72 hours (after Biktarvy®).
Half-life elimination of each of the three active ingredients in Biktarvy® | 0 - 72 hours
  Measurement of half-life elimination of each of the three active ingredients in Biktarvy® (TAF/FTC/BIC), administered in the forms of a complete and solid tablet (phase S), a tablet dissolved in water (phase D) or a tablet crushed and suspended in apple compote (phase C)
  Samples taken at the following times:
  0 hour (right before taking Biktarvy®); 0.5 hour; 1 hours; 1.5 hour; 2 hours; 2.5 hours; 3 hours; 4 hours; 8 hours; 12 hours; 24 hours; 36 hours; 48 hours and 72 hours (after Biktarvy®).
Area Under the curve of each of the three active ingredients in Biktarvy® | 0 - 72 hours
  Measurement of area under the curve of each of the three active ingredients in Biktarvy® (TAF/FTC/BIC), administered in the forms of a complete and solid tablet (phase S), a tablet dissolved in water (phase D) or a tablet crushed and suspended in apple compote (phase C)
  Samples taken at the following times:
  0 hour (right before taking Biktarvy®); 0.5 hour; 1 hours; 1.5 hour; 2 hours; 2.5 hours; 3 hours; 4 hours; 8 hours; 12 hours; 24 hours; 36 hours; 48 hours and 72 hours (after Biktarvy®).

SECONDARY OUTCOMES:
collection of adverse events at all grades | baseline up to 30 days after last administration
  Safety criteria: number and nature of adverse events per patient (all grades (CTCAE scale, version 5.0)), from when the consent form is signed to one month after the last administration of the drug.
tolerance | baseline
  Measuring the tolerance of the three methods of administration (taste, how easy it is to take) by using simple verbal scales graduated 0 to 10.
Volunteer's preference | baseline
  Volunteer's preference by classifying the three methods of administration in order.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France

REFERENCES:
- [Derived] Hocqueloux L, Lefeuvre S, Bois J, Brucato S, Alix A, Valentin C, Peyro-Saint-Paul L, Got L, Fournel F, Dargere S, Prazuck T, Fournier A, Gregoire N, McNicholl I, Parienti JJ. Bioavailability of dissolved and crushed single tablets of bictegravir, emtricitabine, tenofovir alafenamide in healthy adults: the SOLUBIC randomized crossover study. J Antimicrob Chemother. 2022 Dec 23;78(1):161-168. doi: 10.1093/jac/dkac369. PMID 36322475